CLINICAL TRIAL: NCT02708745
Title: Use of a Novel Parent-Report Measure to Improve Childhood Vaccine Uptake: The Screening for Hesitancy to Optimize Talk (SHOT) Study
Brief Title: Screening for Hesitancy to Optimize Talk
Acronym: SHOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Kaiser Permanente (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Douglas Opel, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1R21HD083770-01A1 (NIH)
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Preventive Health Services
Keywords: communication; immunization
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Parent participants will receive a placebo survey about their attitudes toward common child health topics before their child's health supervision visit.
  Interventions: Behavioral: Placebo Survey
- Intervention Arm (Experimental): Parent participants will also receive the intervention survey about their attitudes toward childhood vaccines before their child's health supervision visit.
  Interventions: Behavioral: Intervention Survey

INTERVENTIONS:
Behavioral: Intervention Survey
  Arms: Intervention Arm
Behavioral: Placebo Survey
  Arms: Placebo Arm

SUMMARY:
The overall goal of this project is to determine whether integrating a novel parent-report measure of vaccine hesitancy into pediatric primary care is effective in improving acceptance of childhood vaccines among vaccine-hesitant parents.

DETAILED DESCRIPTION:
The primary goal of this project is to evaluate the effectiveness of an innovative intervention designed to address these barriers-the Screening for Hesitancy to Optimize Talk (SHOT) intervention-in improving provider-parent vaccine discussions and increasing vaccine acceptance. The SHOT intervention involves administering a validated parent-report measure to parents and communicating their score and item-specific responses to their child's provider before their child's 2 and 6 month health supervision visits. The survey contains 15 questions regarding Health Belief Model concepts that influence parent vaccination behavior and has been shown to predict under-immunization.

Our specific aims are to (1) evaluate the impact of the SHOT intervention on a child's immunization status using a matched-pair, cluster randomized controlled trial design; (2) assess how parents' ratings of their vaccine discussions with their child's provider change as a function of the SHOT intervention; and (3) compare pre- and post-study perceptions of barriers to quality vaccine discussions with parents between providers in the SHOT and control arm.

ELIGIBILITY:
Inclusion Criteria:

Parents: Parents must be English speaking, ≥18 years old, have a newborn singleton infant ≤2 months, born at ≥35 weeks gestation who is receiving pediatric care at an enrolled Kaiser Permanente or Allegro Pediatrics clinic, and be vaccine hesitant (defined as positive screening score on eligibility survey).

Newborns: Newborns 0 - 2 months old whose parents enroll in the study will be invited to participate.

Providers: All pediatric and family practice providers at Kaiser Permanente and Allegro Pediatrics primary clinics within a 5 county region in western Washington (Snohomish, King, Pierce, Thurston, and Kitsap Counties) will be eligible to participate.

Exclusion Criteria:

Parents/Children: Parents who are not 18 years or older, require language interpretation for medical care, have an infant born <35 weeks gestation, are not vaccine hesitant or will not be taking their child to a participating clinic for health supervision visits will be excluded.

Providers: Clinics and providers outside the 5 county region in western Washington (Snohomish, King, Pierce, Thurston, and Kitsap) will be excluded.

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2016-03; Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Opel, MD, MPH, Principal Investigator — Seattle Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammer LD, Curry ES, Harlor AD, Laughlin JJ, Leeds AJ, Lessin HR, Rodgers CT, Granado-Villar DC, Brown JM, Cotton WH, Gaines BM, Gambon TB, Gitterman BA, Gorski PA, Kraft CA, Marino RV, Paz-Soldan GJ, Zind B; Committee on Practice and Ambulatory Medicine; Council on Community Pediatrics. Increasing immunization coverage. Pediatrics. 2010 Jun;125(6):1295-304. doi: 10.1542/peds.2010-0743. Epub 2010 May 31. PMID 20513736
- [Background] Opel DJ, Heritage J, Taylor JA, Mangione-Smith R, Salas HS, Devere V, Zhou C, Robinson JD. The architecture of provider-parent vaccine discussions at health supervision visits. Pediatrics. 2013 Dec;132(6):1037-46. doi: 10.1542/peds.2013-2037. Epub 2013 Nov 4. PMID 24190677
- [Background] Healy CM, Montesinos DP, Middleman AB. Parent and provider perspectives on immunization: are providers overestimating parental concerns? Vaccine. 2014 Jan 23;32(5):579-84. doi: 10.1016/j.vaccine.2013.11.076. Epub 2013 Dec 4. PMID 24315883
- [Background] McCauley MM, Kennedy A, Basket M, Sheedy K. Exploring the choice to refuse or delay vaccines: a national survey of parents of 6- through 23-month-olds. Acad Pediatr. 2012 Sep-Oct;12(5):375-83. doi: 10.1016/j.acap.2012.06.007. Epub 2012 Aug 22. PMID 22921495
- [Background] Opel DJ, Mangione-Smith R, Taylor JA, Korfiatis C, Wiese C, Catz S, Martin DP. Development of a survey to identify vaccine-hesitant parents: the parent attitudes about childhood vaccines survey. Hum Vaccin. 2011 Apr;7(4):419-25. doi: 10.4161/hv.7.4.14120. Epub 2011 Apr 1. PMID 21389777
- [Background] Opel DJ, Taylor JA, Mangione-Smith R, Solomon C, Zhao C, Catz S, Martin D. Validity and reliability of a survey to identify vaccine-hesitant parents. Vaccine. 2011 Sep 2;29(38):6598-605. doi: 10.1016/j.vaccine.2011.06.115. Epub 2011 Jul 16. PMID 21763384
- [Background] Opel DJ, Taylor JA, Zhou C, Catz S, Myaing M, Mangione-Smith R. The relationship between parent attitudes about childhood vaccines survey scores and future child immunization status: a validation study. JAMA Pediatr. 2013 Nov;167(11):1065-71. doi: 10.1001/jamapediatrics.2013.2483. PMID 24061681
- [Derived] Opel DJ, Henrikson N, Lepere K, Hawkes R, Zhou C, Dunn J, Taylor JA. Previsit Screening for Parental Vaccine Hesitancy: A Cluster Randomized Trial. Pediatrics. 2019 Nov;144(5):e20190802. doi: 10.1542/peds.2019-0802. Epub 2019 Oct 9. PMID 31597690

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: Parent participants will receive a placebo survey about their attitudes toward common child health topics before their child's health supervision visit.
  Placebo Survey
- Intervention Arm: Parent participants will also receive the intervention survey about their attitudes toward childhood vaccines before their child's health supervision visit.
  Intervention Survey
- Pre-Intervention Providers: Providers at enrolled clinics who completed a survey before the parent-level intervention period
- Post-Intervention Providers: Providers at enrolled clinics who completed a survey after the parent-level intervention period
Period: Overall Study
Arm/Group | Placebo Arm | Intervention Arm | Pre-Intervention Providers | Post-Intervention Providers
Started | 91 | 69 | 204 | 198
Completed | 91 | 65 | 121 | 116
Not Completed | 0 | 4 | 83 | 82

BASELINE CHARACTERISTICS:
Population: In 'placebo arm' and 'intervention arm': parent/child dyads; In 'pre-intervention providers' group: providers at enrolled clinics who completed a survey before the parent-level intervention; In 'post-intervention providers' group: providers at enrolled clinics who completed a survey after the parent-level intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Intervention Arm | Pre-Intervention Providers | Post-Intervention Providers | Total
Number analyzed (Participants) | 91 | 65 | 121 | 116 | 393
Age, Categorical [Count of Participants; unit: Participants] — Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    <=18 years | 0 | 0 |  |  | 0
    Between 18 and 65 years | 91 | 65 |  |  | 156
    >=65 years | 0 | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There was missing data from providers on this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 120 | 113 | 389
    Female | 61 | 41 | 84 | 82 | 268
    Male | 30 | 24 | 36 | 31 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 3 | 3 | 15
  Not Hispanic or Latino | 79 | 58 | 117 | 108 | 362
  Unknown or Not Reported | 8 | 2 | 1 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 25 | 14 | 23 | 26 | 88
  Native Hawaiian or Other Pacific Islander | 7 | 7 | 0 | 0 | 14
  Black or African American | 0 | 0 | 5 | 4 | 9
  White | 43 | 35 | 85 | 80 | 243
  More than one race | 6 | 8 | 6 | 3 | 23
  Unknown or Not Reported | 10 | 1 | 2 | 3 | 16
Number of parent participants married or living with a partner [Count of Participants; unit: Participants] — Married or living with a partner Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    (all) | 79 | 59 |  |  | 138
Number of parent participants with a level of education greater than or equal to 4 years of college [Count of Participants; unit: Participants] — greater than or equal to 4 years of college Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    (all) | 66 | 45 |  |  | 111
Number of parent participants with a household income of greater than $75,000 per year [Count of Participants; unit: Participants] — greater than $75,000 per year Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    (all) | 53 | 43 |  |  | 96
Number of parent participants who were mothers [Count of Participants; unit: Participants] — mother Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    (all) | 61 | 41 |  |  | 102
Number of parent participants who had 1 child in the household [Count of Participants; unit: Participants] — 1 Child in Household Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    (all) | 37 | 38 |  |  | 75
PACV-4 Score [Count of Participants; unit: Participants] — The PACV-4 is a 4-item survey to identify vaccine-hesitant parents. The 4 items are 1) Have you ever delayed having your child get a shot for reasons other than illness or allergy?; 2) How concerned are you that a shot might not prevent the disease?; 3) Overall, how hesitant about childhood shots would you consider yourself to be?; and 4) I trust the information I receive about shots. The PACV-4 is scored from 1-4, with the hesitant response for each item (e.g. the 'yes' response to item 1) receiving a numeric score of 1. A parent was eligible for the study if they scored 2 or higher. Population: Data was not collected from providers for this measure
  Participants
    number analyzed (Participants) | 91 | 65 | 0 | 0 | 156
    2 | 45 | 27 |  |  | 72
    3 | 28 | 23 |  |  | 51
    4 | 17 | 13 |  |  | 30
    missing | 1 | 2 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Child's Mean Percent Days Under-immunized
Description: Mean percent days under-immunized among children of parents who received (vs. did not receive) the intervention
Time Frame: Child's immunization status at 8 months of age
Population: Mean percent days under-immunized of child participants by study arm
Measure: Mean (95% Confidence Interval); unit: percentage of days under-immunized
Arm/Group | Placebo Arm | Intervention Arm
Number analyzed (Participants) | 91 | 65
percentage of days under-immunized | 19.1 [12 to 26.3] | 25.2 [16 to 34.5]
Statistical Analysis 1: Comparison: Placebo Arm vs Intervention Arm; Test type: Superiority; p = .29, t-test, 2 sided

2. Secondary Outcome: Number of Parents With a Highly Rated Visit Experience
Description: Score on a 15-item parent-completed visit experience survey (minimum score 15; maximum score 105, with higher scores suggesting a higher rated visit experience)
Time Frame: 24-48 hours after the 6 month health supervision visit
Population: Proportion of parents with a highly-rated visit experience by study arm, defined as those who scored 90 or higher (out of 105) on the visit experience survey
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Parents in this arm received the intervention
- Placebo: Parents in this arm did not receive the intervention
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 65 | 91
Participants | 44 | 52
Statistical Analysis 1: Comparison: Experimental vs Placebo; Test type: Superiority; p = 0.18, Chi-squared

3. Secondary Outcome: Provider Perceptions of Barriers to the Vaccine Discussion
Description: Provider-reported ratings of the significance of 3 barriers to the vaccine discussion: a) not having enough time to discuss parental vaccine concerns, b) not realizing until late in the visit that a parent had vaccine concerns, and c) not understanding a parent's specific vaccine concerns to be barriers pre- and post-intervention
Time Frame: Change post-intervention from pre-intervention
Population: Proportion in arm who rated barrier as significant (3-5 on a 1-5 scale, where 1=not at all significant and 5=very significant)
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Intervention Providers: Providers rated the significance of the 3 barriers to the vaccine discussion before the parent-level intervention period
- Post-Intervention Providers: Providers rated the significance of the 3 barriers to the vaccine discussion after the parent-level intervention period
Arm/Group | Pre-Intervention Providers | Post-Intervention Providers
Number analyzed (Participants) | 121 | 116
Participants
  Barrier: Not having enough time: number analyzed (Participants) | 62 | 11
  Barrier: Not having enough time: Placebo Arm | 31 | 6
  Barrier: Not having enough time: Intervention Arm | 31 | 5
  Barrier: Not realizing until late in the visit: number analyzed (Participants) | 53 | 14
  Barrier: Not realizing until late in the visit: Placebo Arm | 26 | 9
  Barrier: Not realizing until late in the visit: Intervention Arm | 27 | 5
  Barrier: Not understanding a parent's concerns: number analyzed (Participants) | 53 | 11
  Barrier: Not understanding a parent's concerns: Placebo Arm | 25 | 6
  Barrier: Not understanding a parent's concerns: Intervention Arm | 28 | 5
Statistical Analysis 1: Comparison: Pre-Intervention Providers vs Post-Intervention Providers; Test type: Superiority; p = 0.78, Chi-squared — For the barrier 'not having enough time to discuss vaccine concerns', P=0.78. For the barrier 'not realizing until late in visit that parent had vaccine concerns', P=0.37. For the barrier 'not understanding parent specific vaccine concerns', P=0.66

ADVERSE EVENTS:
Time Frame: 2 years 1 month
Description: No adverse events occurred
Arm/Group | Placebo Arm | Intervention Arm | Pre-Intervention Providers | Post-Intervention Providers
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/65 | 0/121 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/65 | 0/121 | 0/116
Other Adverse Events (participants affected / at risk) | 0/91 | 0/65 | 0/121 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02708745/Prot_SAP_000.pdf